CLINICAL TRIAL: NCT00171522
Title: A Randomized, Open-label, Pilot Crossover Study to Assess the Patient Preference of Tegaserod Versus Polyethylene Glycol 3350 in Patients With Constipation
Brief Title: Preference of Tegaserod vs. PEG 3350 in Patients With Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHTF919EUS49
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Constipation
Keywords: Constipation; Tegaserod; Polyethylene Glycol 3350; PEG
MeSH Terms: conditions — Constipation | interventions — tegaserod; polyethylene glycol 3350

INTERVENTIONS:
Drug: Tegaserod and Polyethylene Glycol 3350

SUMMARY:
To determine whether female patients have a preference for tegaserod of PEG 3350 relative to dosage form, convenience, ease of administration and taste

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 64 years of age
* Patients with constipation as defined by the Rome II criteria

Exclusion Criteria:

* Patients who have been previously been treated with tegaserod and/or PEG 3350
* Evidence of cathartic colon or a history of laxative abuse or laxative dependence
* History of fecal impaction which necessitated surgical intervention
* Patients with clinically significant abnormal TSH levels at screening
* Women who are pregnant or breast feeding

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 64 Years | Sex: Female
Age Groups: Adult
Enrollment: 52
Dates: Start 2005-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
To determine after 14 / 35 days of treatment if women with constipation have a preference for tegaserod compared to PEG 3350, based on the assessment of the Constipation Treatment questionnaire (satisfaction with treatment, willingness to re-use)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Harmony Clinical Research, Oro Valley, Arizona
  - Central Phoenix Medical Clinic, LLC, Phoenix, Arizona
  - Adobe Gastroenterology, PC, Tucson, Arizona
  - Associated Pharmaceutical Research Center, Inc, Buena Park, California
  - Clinical Trial Management of Boca Raton, Inc., Boca Raton, Florida
  - Health Science Center, Pratt, Kansas
  - Beth Israel Deacon Medical Center, Boston, Massachusetts
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - MBS Clinical Research, LLC, Margate City, New Jersey
  - Midwest Clinical Research, Bellbrook, Ohio
  - Associates in Gastroenterology, Hermitage, Tennessee
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - National Clinical Research, Inc, Richmond, Virginia
  - East Coast Clinical Research, Virginia Beach, Virginia